CLINICAL TRIAL: NCT00744471
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE HIP.
Brief Title: Tanezumab in Osteoarthritis Of The Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091014; P3 OA HIP (Other: Alias Study Number)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Arthritis; Osteoarthritis; Osteoarthritis, Hip
Keywords: monoclonal antibody RN624 PF-04383119 nerve growth factor anti-nerve growth OA
MeSH Terms: conditions — Arthritis; Osteoarthritis; Osteoarthritis, Hip | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tanezumab 10 mg (Experimental): Tanezumab 10 mg IV every 8 weeks
  Interventions: Biological: tanezumab
- Tanezumab 5 mg (Experimental): Tanezumab 5mg IV every 8 weeks
  Interventions: Biological: tanezumab
- Tanezumab 2.5 mg (Experimental): Tanezumab 2.5 mg IV every 8 weeks.
  Interventions: Biological: tanezumab
- Placebo (Experimental): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: tanezumab — Tanezumab 10 mg IV every 8 weeks
  Arms: Tanezumab 10 mg
Biological: tanezumab — Tanezumab 5mg IV every 8 weeks
  Arms: Tanezumab 5 mg
Biological: tanezumab — Tanezumab 2.5 mg IV every 8 weeks.
  Arms: Tanezumab 2.5 mg
Biological: Placebo — Placebo to match tanezumab IV every 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of 3 doses of tanezumab in osteoarthritis of the hip in patients

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the hip according to ACR criteria with Kellgren-Lawrence x-ray grade of 2
* Unwilling or unable to take non-opiate pain medications, for whom non-opiate pain medications have not provided adequate pain relief or are candidates for Hip injections, arthroplasty or replacement surgery
* Pain level and function levels as required by the protocol at Screening and Baseline
* Willing to discontinue pain medications (acetaminophen will be permitted up to a certain level) before and during the study
* Must agree to the contraceptive requirements of the protocol if applicable
* Must agree to the treatment plan, scheduled visits, and procedures of the protocol

Exclusion Criteria:

* Pregnancy
* BMI greater than 39
* Other severe pain, significant cardiac, neurological or psychological conditions, or above the protocol limits for laboratory and blood pressure results

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2010-03-15 (Actual); Study Completion 2010-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (99):
  - Horizon Research Group, Mobile, Alabama
  - Arizona Arthritis & Rheumatology Associates, PC, Paradise Valley, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Clinical Research Advantage, Inc. /Stonecreek Medical Associates, PC, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, PC, Phoenix, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - St. Joseph's Mercy Clinic, Hot Springs, Arkansas
  - Providence Clinical Research, Burbank, California
  - Arthritis Medical Clinic of North County, Inc., Escondido, California
  - Talbert Medical Group, Huntington Beach, California
  - Trinity Clinical Trials, Santa Ana, California
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Avail Clinical Research, DeLand, Florida
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - International Research Associates, LLC, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Advent Clinical Research Centers, Pinellas Park, Florida
  - Avivoclin Clinical Services, Port Orange, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - All Florida Orthopaedic Associates, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Laureate Clinical Reseach Group, Atlanta, Georgia
  - Early Family Practice Center, Fort Valley, Georgia
  - Northeast Georgia Diagnostic Clinic, Gainesville, Georgia
  - North Georgia Clinical Research, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal medicine, Woodstock, Georgia
  - Sonora Clinical Research, Boise, Idaho
  - The Arthritis Center, Springfield, Illinois
  - American Health Network of IN, LLC, Fishers, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Maine Research Associates, Auburn, Maine
  - The Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Mansfield Health Center, Mansfield, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Ann Arbor Clinical Research, Ann Arbor, Michigan
  - Rheumatology, PC, Kalamazoo, Michigan
  - MAPS Applied Research Center, Edina, Minnesota
  - Medical Advanced Pain Specialists, Edina, Minnesota
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical, Las Vegas, Nevada
  - Office of Dr. Danka Michaels, MD, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Incorporated, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Center of Brooklyn Heights, Brooklyn, New York
  - The Medical Research Network, LLC, New York, New York
  - Prem C. Chatpar, MD, LLC, Plainview, New York
  - Office of Dr. Andrew Porges, Roslyn, New York
  - Carolina Bone & Joint, P.A., Charlotte, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Consultants for Clinical Research/Ohio GI and Liver Institute, Cincinnati, Ohio
  - Hilltop Physicians Inc, Hightop Medical Research Center, Cincinnati, Ohio
  - Southwest Rheumatology and Research Group, LLC, Middleburg Heights, Ohio
  - Pharmacotherapy Research Associates,Inc, Zanesville, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - EPIC Imaging West, Beaverton, Oregon
  - EPIC Imaging East, Portland, Oregon
  - Covance CRU, Inc., Portland, Oregon
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Appalachian Medical Research Inc., Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Capital Medical Clinic, Austin, Texas
  - Walter Chase MD, Austin, Texas
  - Radiant Research, Dallas, Texas
  - Rheumatic Disease Clinical Research Center, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Pioneet Research Solutions, Inc, Houston, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Radiant Research San Antonio NE, San Antonio, Texas
  - Texas Arthritis Research Center, PA, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sushma V. Gorrela, MD, Spring, Texas
  - Optimum Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Internal Medicine Northwest, Frank S Baker Center, Tacoma, Washington
  - Clinical Trials Northwest, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- [Derived] Brown MT, Murphy FT, Radin DM, Davignon I, Smith MD, West CR. Tanezumab reduces osteoarthritic hip pain: results of a randomized, double-blind, placebo-controlled phase III trial. Arthritis Rheum. 2013 Jul;65(7):1795-803. doi: 10.1002/art.37950. PMID 23553790

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion over 5 minutes at Day 1, Week 8 and Week 16.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Started | 156 | 156 | 158 | 157
Treated | 155 | 155 | 154 | 157
Completed | 13 | 11 | 6 | 9
Not Completed | 143 | 145 | 152 | 148
Not completed — Randomized but not treated | 1 | 1 | 4 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Adverse Event | 6 | 7 | 5 | 9
Not completed — Withdrawal by Subject | 9 | 9 | 15 | 12
Not completed — Protocol Violation | 1 | 4 | 1 | 2
Not completed — Entered extension study | 41 | 84 | 100 | 91
Not completed — Other | 2 | 3 | 6 | 2
Not completed — Lack of Efficacy | 83 | 37 | 19 | 31
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous (IV) study medication (either tanezumab or matching placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg | Total
Number analyzed (Participants) | 155 | 155 | 154 | 157 | 621
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 11 | 8 | 11 | 6 | 36
  Between 45 and 64 years | 84 | 86 | 74 | 82 | 326
  >= 65 years | 60 | 61 | 69 | 69 | 259
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 101 | 92 | 88 | 384
  Male | 52 | 54 | 62 | 69 | 237

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in hip joint during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline (Day 1), Week 16
Population: Modified intent-to-treat (mITT) analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. BOCF method used to impute missing values. "Overall Number of participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Baseline | 7.26 (1.39) | 7.20 (1.44) | 7.24 (1.46) | 7.33 (1.64)
  Change at Week 16 | -1.65 (2.44) | -2.86 (2.73) | -3.35 (2.76) | -3.37 (2.80)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 16: Analysis of Covariance (ANCOVA) was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; Least Squares (LS) Mean Difference = -1.28, 95% CI 2-sided [-1.87 to -0.69], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 16: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.69, 95% CI 2-sided [-2.28 to -1.10], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.75, 95% CI 2-sided [-2.34 to -1.16], Standard Error of Mean 0.30

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in hip joint during past 48 hours. It is calculated as mean of the scores from 17 individual questions scored on a NRS of 0 to 10, where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 to 10, where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 16
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site.BOCF method used to impute missing values. "Overall Number of participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Baseline | 6.79 (1.56) | 6.79 (1.63) | 6.82 (1.70) | 6.83 (1.83)
  Change at Week 16 | -1.39 (2.25) | -2.54 (2.72) | -2.88 (2.70) | -2.96 (2.68)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 16: ANCOVA was performed with treatment as main effects, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.18, 95% CI 2-sided [-1.74 to -0.61], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 16: ANCOVA model includes treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.49, 95% CI 2-sided [-2.06 to -0.92], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.61, 95% CI 2-sided [-2.17 to -1.04], Standard Error of Mean 0.29

3. Primary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 16: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways your osteoarthritis in your hip joint affects you, how are you doing today?", participants responded by using a 5-point scale where 1 = very good (no symptom and limitation of normal activities) and 5 = very poor (very severe symptoms and inability to carry out normal activities), where lower scores indicates better condition.
Time Frame: Baseline, Week 16
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. BOCF method used to impute missing values. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Baseline | 3.47 (0.60) | 3.55 (0.62) | 3.51 (0.64) | 3.46 (0.66)
  Change at Week 16 | -0.34 (0.69) | -0.67 (0.87) | -0.80 (1.00) | -0.80 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 16: ANCOVA model includes treatment as main effect, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.32, 95% CI 2-sided [-0.51 to -0.13], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.45, 95% CI 2-sided [-0.64 to -0.25], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.47, 95% CI 2-sided [-0.66 to -0.28], Standard Error of Mean 0.10

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in Pain Subscale Score at Week 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -1.94 (2.08) | -3.32 (2.59) | -3.71 (2.53) | -3.30 (2.52)
  Change at Week 4 | -1.92 (2.17) | -3.46 (2.64) | -3.99 (2.63) | -3.88 (2.74)
  Change at Week 8 | -1.74 (2.33) | -2.76 (2.62) | -3.36 (2.60) | -3.70 (2.71)
  Change at Week 12 | -1.81 (2.44) | -3.24 (2.89) | -3.67 (2.79) | -3.77 (2.98)
  Change at Week 24 | -1.45 (2.43) | -2.54 (2.74) | -3.00 (2.80) | -3.06 (2.80)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 2: ANCOVA model includes treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.41, 95% CI 2-sided [-1.93 to -0.88], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.73, 95% CI 2-sided [-2.26 to -1.20], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.33, 95% CI 2-sided [-1.85 to -0.80], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 4: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.57, 95% CI 2-sided [-2.11 to -1.02], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.03, 95% CI 2-sided [-2.57 to -1.48], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.95, 95% CI 2-sided [-2.50 to -1.41], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 8: ANCOVA model was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.09, 95% CI 2-sided [-1.65 to -0.53], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 8: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.64, 95% CI 2-sided [-2.20 to -1.08], Standard Error of Mean 0.29
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.00, 95% CI 2-sided [-2.56 to -1.45], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 12: ANCOVA model was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.49, 95% CI 2-sided [-2.10 to -0.88], Standard Error of Mean 0.31
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.85, 95% CI 2-sided [-2.46 to -1.25], Standard Error of Mean 0.31
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.97, 95% CI 2-sided [-2.57 to -1.37], Standard Error of Mean 0.31
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 24: ANCOVA model was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.16, 95% CI 2-sided [-1.75 to -0.56], Standard Error of Mean 0.30
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.52, 95% CI 2-sided [-2.12 to -0.92], Standard Error of Mean 0.30
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.60, 95% CI 2-sided [-2.20 to -1.01], Standard Error of Mean 0.30

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in Pain Subscale Score at Week 2, 4, 8, 12,16 and 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. LOCF method used to impute missing values. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -1.94 (2.08) | -3.32 (2.59) | -3.71 (2.53) | -3.30 (2.52)
  Change at Week 4 | -2.02 (2.18) | -3.55 (2.59) | -4.04 (2.60) | -4.04 (2.59)
  Change at Week 8 | -1.86 (2.32) | -2.95 (2.50) | -3.52 (2.61) | -3.89 (2.69)
  Change at Week 12 | -2.12 (2.48) | -3.58 (2.71) | -4.03 (2.67) | -4.35 (2.69)
  Change at Week 16 | -2.05 (2.47) | -3.23 (2.59) | -3.66 (2.74) | -3.96 (2.61)
  Change at Week 24 | -1.97 (2.50) | -3.16 (2.62) | -3.56 (2.74) | -3.77 (2.60)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 2: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.41, 95% CI 2-sided [-1.93 to -0.88], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.73, 95% CI 2-sided [-2.26 to -1.20], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.33, 95% CI 2-sided [-1.85 to -0.80], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.55, 95% CI 2-sided [-2.08 to -1.02], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.99, 95% CI 2-sided [-2.52 to -1.46], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.01, 95% CI 2-sided [-2.54 to -1.48], Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.17, 95% CI 2-sided [-1.71 to -0.63], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.66, 95% CI 2-sided [-2.21 to -1.12], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.06, 95% CI 2-sided [-2.60 to -1.52], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 12: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.55, 95% CI 2-sided [-2.11 to -0.99], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.88, 95% CI 2-sided [-2.45 to -1.32], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.26, 95% CI 2-sided [-2.82 to -1.70], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.27, 95% CI 2-sided [-1.82 to -0.71], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.59, 95% CI 2-sided [-2.15 to -1.03], Standard Error of Mean 0.28
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.96, 95% CI 2-sided [-2.51 to -1.40], Standard Error of Mean 0.28
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 24: ANCOVA was performed with treatment as main effects, baseline value as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.29, 95% CI 2-sided [-1.85 to -0.72], Standard Error of Mean 0.29
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.58, 95% CI 2-sided [-2.15 to -1.01], Standard Error of Mean 0.29
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.83, 95% CI 2-sided [-2.40 to -1.27], Standard Error of Mean 0.29

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Subscale Score at Week 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in hip joint during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -1.56 (2.01) | -2.88 (2.53) | -3.32 (2.50) | -2.90 (2.46)
  Change at Week 4 | -1.44 (1.99) | -3.06 (2.60) | -3.62 (2.43) | -3.40 (2.57)
  Change at Week 8 | -1.33 (2.21) | -2.48 (2.66) | -2.95 (2.45) | -3.17 (2.61)
  Change at Week 12 | -1.52 (2.19) | -2.86 (2.86) | -3.27 (2.71) | -3.39 (2.85)
  Change at Week 24 | -1.27 (2.18) | -2.19 (2.65) | -2.62 (2.61) | -2.78 (2.67)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 2: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.31, 95% CI 2-sided [-1.83 to -0.80], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.71, 95% CI 2-sided [-2.23 to -1.19], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.32, 95% CI 2-sided [-1.83 to -0.80], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 4: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.60, 95% CI 2-sided [-2.12 to -1.08], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.12, 95% CI 2-sided [-2.64 to -1.60], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.94, 95% CI 2-sided [-2.46 to -1.43], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 8: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.18, 95% CI 2-sided [-1.72 to -0.64], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.64, 95% CI 2-sided [-2.18 to -1.09], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.89, 95% CI 2-sided [-2.43 to -1.35], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 12: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.35, 95% CI 2-sided [-1.93 to -0.77], Standard Error of Mean 0.30
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 12 :Analysis of Covariance (ANCOVA) was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean difference = -1.73, 95% CI 2-sided [-2.31 to -1.15], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.89, 95% CI 2-sided [-2.47 to -1.32], Standard Error of Mean 0.29
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 24 : ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.96, 95% CI 2-sided [-1.52 to -0.40], Standard Error of Mean 0.29
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; Change at Week 24 :Analysis of Covariance (ANCOVA) was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.35, 95% CI 2-sided [-1.91 to -0.78], Standard Error of Mean 0.29
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 14]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.53, 95% CI 2-sided [-2.09 to -0.97], Standard Error of Mean 0.28

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Subscale at Week 2, 4, 8, 12, 16 and 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. LOCF method used to impute missing values. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -1.56 (2.01) | -2.88 (2.53) | -3.32 (2.50) | -2.90 (2.46)
  Change at Week 4 | -1.51 (2.05) | -3.13 (2.59) | -3.67 (2.43) | -3.52 (2.48)
  Change at Week 8 | -1.40 (2.24) | -2.66 (2.64) | -3.14 (2.44) | -3.35 (2.64)
  Change at Week 12 | -1.61 (2.39) | -3.12 (2.82) | -3.58 (2.63) | -3.85 (2.68)
  Change at Week 16 | -1.56 (2.41) | -2.83 (2.72) | -3.16 (2.72) | -3.42 (2.60)
  Change at Week 24 | -1.46 (2.42) | -2.71 (2.71) | -3.09 (2.61) | -3.34 (2.56)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.31, 95% CI 2-sided [-1.83 to -0.80], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.71, 95% CI 2-sided [-2.23 to -1.19], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.32, 95% CI 2-sided [-1.83 to -0.80], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.59, 95% CI 2-sided [-2.10 to -1.08], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.10, 95% CI 2-sided [-2.61 to -1.59], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.00, 95% CI 2-sided [-2.51 to -1.49], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.29, 95% CI 2-sided [-1.83 to -0.76], Standard Error of Mean 0.27
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.72, 95% CI 2-sided [-2.26 to -1.19], Standard Error of Mean 0.27
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; Slope = -1.99, 95% CI 2-sided [-2.53 to -1.46], Standard Error of Mean 0.27
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.56, 95% CI 2-sided [-2.11 to -1.00], Standard Error of Mean 0.28
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean difference = -1.93, 95% CI 2-sided [-2.49 to -1.37], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -2.28, 95% CI 2-sided [-2.83 to -1.72], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 16: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.31, 95% CI 2-sided [-1.87 to -0.75], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.58, 95% CI 2-sided [-2.14 to -1.02], Standard Error of Mean 0.29
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.92, 95% CI 2-sided [-2.47 to -1.36], Standard Error of Mean 0.28
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; Change at Week 24: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.30, 95% CI 2-sided [-1.86 to -0.74], Standard Error of Mean 0.28
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -1.61, 95% CI 2-sided [-2.17 to -1.05], Standard Error of Mean 0.28
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; Slope = -1.91, 95% CI 2-sided [-2.47 to -1.36], Standard Error of Mean 0.28

8. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -0.41 (0.83) | -0.83 (0.94) | -1.08 (1.02) | -0.81 (0.92)
  Change at Week 4 | -0.44 (0.79) | -0.93 (0.88) | -1.16 (0.96) | -0.97 (0.98)
  Change at Week 8 | -0.43 (0.86) | -0.65 (0.93) | -0.93 (1.03) | -0.86 (0.94)
  Change at Week 12 | -0.41 (0.76) | -0.78 (0.93) | -1.03 (1.05) | -0.92 (0.96)
  Change at Week 24 | -0.36 (0.72) | -0.61 (0.84) | -0.78 (1.00) | -0.60 (0.89)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.37, 95% CI 2-sided [-0.55 to -0.18], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.64, 95% CI 2-sided [-0.83 to -0.45], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.60 to -0.22], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.65 to -0.27], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.69, 95% CI 2-sided [-0.88 to -0.50], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.55, 95% CI 2-sided [-0.73 to -0.36], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.054, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.19, 95% CI 2-sided [-0.39 to 0.00], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.48, 95% CI 2-sided [-0.68 to -0.29], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.45, 95% CI 2-sided [-0.65 to -0.26], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.35, 95% CI 2-sided [-0.55 to -0.15], Standard Error of Mean 0.10
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.61, 95% CI 2-sided [-0.81 to -0.40], Standard Error of Mean 0.10
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.53, 95% CI 2-sided [-0.73 to -0.32], Standard Error of Mean 0.10
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.26, 95% CI 2-sided [-0.45 to -0.07], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.60 to -0.22], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.24, 95% CI 2-sided [-0.43 to -0.05], Standard Error of Mean 0.10

9. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12, 16 and 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 150 | 150 | 155
Units on a scale
  Change at Week 2 | -0.41 (0.83) | -0.83 (0.94) | -1.08 (1.02) | -0.81 (0.92)
  Change at Week 4 | -0.45 (0.81) | -0.95 (0.88) | -1.17 (0.97) | -1.03 (0.99)
  Change at Week 8 | -0.46 (0.90) | -0.73 (0.95) | -0.96 (1.04) | -0.90 (0.96)
  Change at Week 12 | -0.44 (0.90) | -0.87 (0.99) | -1.14 (1.05) | -1.01 (1.00)
  Change at Week 16 | -0.38 (0.86) | -0.76 (0.95) | -0.89 (1.05) | -0.88 (0.99)
  Change at Week 24 | -0.42 (0.90) | -0.71 (0.95) | -0.90 (1.08) | -0.74 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.37, 95% CI 2-sided [-0.55 to -0.18], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.64, 95% CI 2-sided [-0.83 to -0.45], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.60 to -0.22], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.65 to -0.27], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.68, 95% CI 2-sided [-0.87 to -0.50], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.58, 95% CI 2-sided [-0.76 to -0.39], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p = 0.022, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.23, 95% CI 2-sided [-0.43 to -0.03], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; Week 8: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.47, 95% CI 2-sided [-0.67 to -0.27], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.65 to -0.26], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.40, 95% CI 2-sided [-0.60 to -0.19], Standard Error of Mean 0.10
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; Week 12: ANCOVA was performed with treatment as main effect, baseline value, as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.68, 95% CI 2-sided [-0.88 to -0.47], Standard Error of Mean 0.10
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.59, 95% CI 2-sided [-0.79 to -0.39], Standard Error of Mean 0.10
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.33, 95% CI 2-sided [-0.53 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.48, 95% CI 2-sided [-0.68 to -0.28], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.51, 95% CI 2-sided [-0.71 to -0.32], Standard Error of Mean 0.10
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.27, 95% CI 2-sided [-0.47 to -0.06], Standard Error of Mean 0.10
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.66 to -0.25], Standard Error of Mean 0.10
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 7, analysis 16]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is based on ANCOVA from pairwise comparisons; LS Mean Difference = -0.33, 95% CI 2-sided [-0.53 to -0.13], Standard Error of Mean 0.10

10. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response: Baseline Observation Carried Forward (BOCF)
Description: A participant was considered as an OMERACT-OARSI responder if at least one of the following criteria were met: Improvement in WOMAC pain or physical function subscale from baseline to week of interest was greater than or equal to (>=) 50 percent (%)and absolute change of >=2 units from baseline at the week of interest, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at the week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis. Score range for PGA: 1 = very good to 5 = very poor, where higher scores=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0 [no pain] to 10 [worst possible pain], higher score=higher pain/difficulty).
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. BOCF method used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2 | 45.5 | 68.7 | 80.0 | 67.7
  Week 4 | 45.5 | 71.3 | 79.3 | 74.8
  Week 8 | 43.5 | 60.7 | 70.7 | 71.0
  Week 12 | 39.6 | 63.3 | 70.0 | 66.5
  Week 16 | 35.1 | 57.3 | 65.3 | 65.8
  Week 24 | 30.5 | 50.7 | 62.0 | 58.7

11. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response: Last Observation Carried Forward (LOCF)
Description: as for outcome 10
Time Frame: Week 2, 4, 8, 12 ,16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. LOCF method used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2 | 45.5 | 68.7 | 80.0 | 67.7
  Week 4 | 48.1 | 73.3 | 81.3 | 78.7
  Week 8 | 47.4 | 66.7 | 75.3 | 75.5
  Week 12 | 50.0 | 74.0 | 78.0 | 78.1
  Week 16 | 48.1 | 68.7 | 72.0 | 77.4
  Week 24 | 46.1 | 66.7 | 73.3 | 74.2

12. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%), and 50 % Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 2, 4, 8, 12, 16, 24: Baseline Observation Carried Forward
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in hip joint during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants with >=30% or >=50% reduction in WOMAC pain subscale score from baseline to specified weeks were reported.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2: >=30% reduction | 38.3 | 64.2 | 70.7 | 58.3
  Week 2: >=50% reduction | 26.0 | 49.0 | 50.7 | 44.2
  Week 4: >=30% reduction | 37.7 | 65.6 | 72.0 | 70.5
  Week 4: >=50% reduction | 23.4 | 50.3 | 59.3 | 56.4
  Week 8: >=30% reduction | 36.4 | 59.6 | 66.0 | 68.4
  Week 8: >= 50% reduction | 22.1 | 40.4 | 48.7 | 52.9
  Week 12: >= 30% reduction | 37.7 | 59.6 | 65.3 | 64.7
  Week 12: >= 50% reduction | 26.0 | 49.0 | 53.3 | 59.0
  Week 16: >= 30% reduction | 32.5 | 56.3 | 63.3 | 61.5
  Week 16: >= 50% reduction | 26.0 | 39.7 | 50.7 | 46.2
  Week 24: >= 30% reduction | 27.9 | 47.7 | 57.3 | 57.1
  Week 24: >= 50% reduction | 19.5 | 37.1 | 46.0 | 44.2

13. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%), and 50% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in hip joint during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a NRS of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Percentage of participants with >=30% or >=50% reduction in WOMAC pain subscale score from baseline to specified weeks were reported.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded and from site 1021. LOCF method was used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2 >= 30% Reduction | 38.3 | 64.2 | 70.7 | 58.3
  Week 2 >= 50% Reduction | 26.0 | 49.0 | 50.7 | 44.2
  Week 4 >= 30% Reduction | 39.0 | 66.9 | 74.0 | 73.7
  Week 4 >= 50% Reduction | 24.7 | 51.7 | 59.3 | 57.7
  Week 8 >= 30% Reduction | 38.3 | 63.6 | 69.3 | 71.8
  Week 8 >= 50% Reduction | 22.7 | 41.1 | 50.0 | 54.5
  Week 12 >= 30% Reduction | 44.8 | 67.5 | 72.7 | 75.6
  Week 12 >= 50% Reduction | 27.9 | 52.3 | 58.0 | 66.0
  Week 16 >= 30% Reduction | 41.6 | 64.9 | 69.3 | 72.4
  Week 16 >= 50% Reduction | 28.6 | 43.7 | 54.7 | 53.2
  Week 24 >= 30% Reduction | 39.6 | 60.9 | 68.0 | 71.2
  Week 24 >= 50% Reduction | 23.4 | 43.7 | 52.7 | 51.9

14. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12 ,16 and 24: Baseline Observation Carried Forward (BOCF)
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?", participants responded by using a 5-point scale where 1 = very good and 5 = very poor where lower scores indicating better condition. Percentage of participants with an improvement of greater than or equal to 2 points from baseline at specified weeks were reported.
Time Frame: Baseline, Week 2, 4, 8, 12 ,16, 24
Population: mITT analysis set: all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. BOCF method was used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2 | 9.7 | 24.0 | 32.0 | 24.5
  Week 4 | 10.4 | 25.3 | 34.0 | 31.6
  Week 8 | 10.4 | 15.3 | 27.3 | 27.1
  Week 12 | 11.7 | 22.0 | 28.7 | 29.7
  Week 16 | 7.1 | 14.7 | 20.0 | 27.7
  Week 24 | 8.4 | 15.3 | 20.7 | 18.7

15. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8, 12, 16, 24: Last Observation Carried Forward (LOCF)
Description: as for outcome 14
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. LOCF method was used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2 | 9.7 | 24.0 | 32.0 | 24.5
  Week 4 | 10.4 | 26.0 | 34.7 | 34.2
  Week 8 | 11.0 | 18.0 | 28.0 | 28.4
  Week 12 | 12.3 | 25.3 | 31.3 | 32.9
  Week 16 | 8.4 | 18.7 | 23.3 | 30.3
  Week 24 | 9.7 | 19.3 | 25.3 | 23.2

16. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in hip joint during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a NRS of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline at Week 16 were reported.
Time Frame: Baseline, Week 16
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. BOCF method was used to impute missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Greater than (>) 0% | 44.8 | 68.2 | 78.7 | 72.4
  >=10% | 40.9 | 64.9 | 73.3 | 70.5
  >=20% | 36.4 | 58.9 | 66.7 | 67.3
  >=30% | 32.5 | 56.3 | 63.3 | 61.5
  >=40% | 29.2 | 50.3 | 54.7 | 53.2
  >=50% | 26.0 | 39.7 | 50.7 | 46.2
  >=60% | 19.5 | 35.8 | 43.3 | 39.7
  >=70% | 13.6 | 28.5 | 36.7 | 35.3
  >=80% | 11.0 | 21.9 | 25.3 | 30.1
  >=90% | 4.5 | 13.2 | 18.0 | 20.5

17. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  >0% | 79.2 | 87.4 | 89.3 | 93.6
  >=10% | 63.6 | 81.5 | 82.0 | 89.7
  >=20% | 50.6 | 70.2 | 74.7 | 81.4
  >=30% | 41.6 | 64.9 | 69.3 | 72.4
  >=40% | 34.4 | 57.0 | 59.3 | 61.5
  >=50% | 28.6 | 43.7 | 54.7 | 53.2
  >=60% | 21.4 | 37.7 | 47.3 | 45.5
  >=70% | 14.3 | 29.1 | 40.7 | 40.4
  >=80% | 11.0 | 21.9 | 28.0 | 34.6
  >=90% | 4.5 | 13.2 | 20.0 | 23.1

18. Secondary Outcome: Change From Baseline in Average Daily Pain Score in the Hip Joint at Week 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: Participants assessed daily average hip joint pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst pain). Post baseline weekly scores were calculated as the mean of the scores over the last 7 days prior to each assessment time point.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline | 6.61 (1.86) | 6.44 (1.89) | 6.71 (1.93) | 6.55 (1.96)
  Change at Week 2 | -1.24 (1.97) | -1.89 (2.40) | -2.51 (2.51) | -2.03 (2.57)
  Change at Week 4 | -1.16 (2.07) | -2.44 (2.42) | -3.10 (2.55) | -2.65 (2.65)
  Change at Week 8 | -0.99 (2.00) | -2.00 (2.37) | -2.50 (2.48) | -2.44 (2.59)
  Change at Week 12 | -1.34 (2.15) | -2.19 (2.58) | -2.84 (2.62) | -2.83 (2.82)
  Change at Week 16 | -1.18 (2.06) | -2.02 (2.40) | -2.39 (2.55) | -2.56 (2.64)
  Change at Week 24 | -0.97 (1.90) | -1.55 (2.29) | -2.24 (2.61) | -2.12 (2.59)

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Week 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in hip joint during past 48 hours. It is calculated as mean of the scores from 2 individual questions each scored on numerical rating scale of 0 (minimum stiffness) to 10 (maximum stiffness), giving an overall possible mean score range of 0 (minimum stiffness) to 10 (maximum stiffness). Higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of hip joint.
Time Frame: Baseline, Week 2, 4, 8, 12 ,16, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline | 7.18 (1.65) | 7.17 (1.69) | 7.02 (2.01) | 7.23 (1.96)
  Change at Week 2 | -1.69 (2.25) | -3.13 (2.67) | -3.47 (3.02) | -3.32 (3.04)
  Change at Week 4 | -1.51 (2.25) | -3.29 (2.72) | -3.80 (2.89) | -3.82 (3.00)
  Change at Week 8 | -1.34 (2.41) | -2.61 (2.69) | -3.17 (3.08) | -3.46 (2.97)
  Change at Week 12 | -1.52 (2.30) | -3.05 (2.95) | -3.60 (3.13) | -3.78 (3.19)
  Change at Week 16 | -1.39 (2.32) | -2.54 (2.76) | -3.09 (3.00) | -3.33 (2.99)
  Change at Week 24 | -1.32 (2.35) | -2.30 (2.77) | -2.93 (3.08) | -3.16 (3.04)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) Average Score at Week 2, 4, 8, 12,16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of hip joint. Each item is scored on a 0 (no pain) to 10 (worst possible pain) NRS scale, where higher scores indicate higher pain/stiffness or worse function. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 (no pain) to 10 (worst possible pain), where higher score indicates worse response.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline | 7.08 (1.39) | 7.05 (1.42) | 7.03 (1.57) | 7.13 (1.63)
  Change at Week 2 | -1.73 (1.97) | -3.13 (2.50) | -3.50 (2.57) | -3.17 (2.55)
  Change at Week 4 | -1.62 (2.02) | -3.27 (2.54) | -3.80 (2.53) | -3.70 (2.65)
  Change at Week 8 | -1.47 (2.22) | -2.63 (2.56) | -3.17 (2.57) | -3.45 (2.66)
  Change at Week 12 | -1.62 (2.23) | -3.05 (2.82) | -3.51 (2.78) | -3.65 (2.93)
  Change at Week 16 | -1.48 (2.28) | -2.65 (2.65) | -3.10 (2.72) | -3.22 (2.73)
  Change at Week 24 | -1.35 (2.28) | -2.34 (2.66) | -2.85 (2.72) | -3.00 (2.72)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) Pain Subscale Item (Pain When Walking on Flat Surface) Score at Week 2, 4, 8, 12, 16 and 24 : Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Participants answered "How much pain have you had when walking on a flat surface?". Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 =extreme pain. Higher scores indicated more pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline | 7.26 (1.66) | 7.21 (1.65) | 7.25 (1.61) | 7.32 (1.76)
  Change at Week 2 | -1.83 (2.39) | -3.31 (2.81) | -3.79 (2.71) | -3.33 (2.54)
  Change at Week 4 | -1.96 (2.38) | -3.40 (2.73) | -4.01 (2.83) | -3.75 (2.87)
  Change at Week 8 | -1.71 (2.55) | -2.84 (2.73) | -3.25 (2.77) | -3.45 (2.71)
  Change at Week 12 | -1.76 (2.51) | -3.13 (2.97) | -3.65 (2.90) | -3.59 (2.96)
  Change at Week 16 | -1.56 (2.43) | -2.73 (2.91) | -3.29 (2.98) | -3.21 (2.81)
  Change at Week 24 | -1.44 (2.43) | -2.45 (2.78) | -2.95 (2.93) | -2.94 (2.80)

22. Secondary Outcome: Change From Baseline of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale (Pain When Going up or Down Stairs) Score at Week 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis. Participants answered "How much pain have you had when going up or down the stairs?". Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = worst possible pain, where higher scores indicating higher pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline | 7.99 (1.46) | 7.94 (1.51) | 7.83 (1.59) | 7.89 (1.81)
  Change at Week 2 | -1.88 (2.15) | -3.42 (2.62) | -3.89 (2.85) | -3.35 (2.71)
  Change at Week 4 | -1.84 (2.26) | -3.59 (2.82) | -4.11 (2.87) | -3.82 (3.03)
  Change at Week 8 | -1.64 (2.32) | -2.87 (2.84) | -3.46 (2.92) | -3.59 (3.05)
  Change at Week 12 | -1.75 (2.49) | -3.39 (3.10) | -3.80 (3.08) | -3.72 (3.23)
  Change at Week 16 | -1.56 (2.50) | -2.95 (3.00) | -3.41 (3.11) | -3.21 (3.03)
  Change at Week 24 | -1.45 (2.46) | -2.54 (2.92) | -2.98 (3.04) | -2.92 (3.03)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: The SF-36 health survey was a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional, domain 8= mental health. Total score for each domain are scaled 0 (minimum) to 100 (maximum), where higher score indicates highest level of functioning.
Time Frame: Baseline, Week 12, 24
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. BOCF method was used to impute missing values. Here, 'Number Analyzed', signified number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Units on a scale
  Baseline: General health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: General health | 64.81 (18.81) | 67.04 (18.12) | 63.74 (18.60) | 64.26 (19.29)
  Baseline: Physical Function: number analyzed (Participants) | 153 | 150 | 150 | 155
  Baseline: Physical Function | 30.56 (19.51) | 29.66 (20.35) | 30.78 (19.69) | 29.48 (19.29)
  Baseline: Role Physical: number analyzed (Participants) | 154 | 150 | 150 | 154
  Baseline: Role Physical | 39.25 (24.74) | 36.96 (24.78) | 38.83 (25.33) | 38.47 (23.86)
  Baseline: Bodily Pain: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: Bodily Pain | 29.70 (13.96) | 29.66 (14.56) | 29.73 (15.78) | 31.25 (16.27)
  Baseline: Vitality: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: Vitality | 47.28 (21.28) | 49.42 (20.93) | 48.04 (20.70) | 46.85 (22.81)
  Baseline: Social Function: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: Social Function | 64.37 (27.11) | 66.67 (25.32) | 63.67 (28.76) | 66.61 (28.39)
  Baseline: Role Emotional: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: Role Emotional | 63.47 (30.57) | 68.94 (28.34) | 67.22 (30.86) | 68.76 (30.26)
  Baseline: Mental Health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Baseline: Mental Health | 72.63 (18.70) | 74.30 (17.76) | 73.90 (18.80) | 73.32 (19.63)
  Change at Week 12:General health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12:General health | 2.07 (9.34) | 4.01 (12.61) | 8.03 (14.24) | 5.27 (13.14)
  Change at Week12:Physical Function: number analyzed (Participants) | 153 | 150 | 150 | 155
  Change at Week12:Physical Function | 6.01 (15.12) | 15.01 (21.38) | 18.52 (25.16) | 18.91 (24.96)
  Change at Week 12: Role Physical: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12: Role Physical | 7.67 (20.91) | 16.88 (23.77) | 22.83 (28.70) | 18.99 (27.10)
  Change at Week 12: Bodily Pain: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12: Bodily Pain | 10.42 (17.62) | 17.97 (22.08) | 25.23 (25.48) | 22.87 (26.10)
  Change at Week 12: Vitality: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12: Vitality | 5.24 (14.14) | 8.13 (15.66) | 10.79 (19.82) | 7.86 (20.03)
  Change at Week 12:Social Function: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12:Social Function | 5.52 (18.91) | 10.25 (22.16) | 12.08 (24.89) | 10.08 (24.88)
  Change at Week 12:Role emotional: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12:Role emotional | 4.44 (21.01) | 8.33 (19.14) | 11.72 (26.93) | 9.68 (23.43)
  Change at Week 12: Mental Health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 12: Mental Health | 3.77 (11.86) | 4.07 (13.44) | 5.73 (15.87) | 2.55 (16.15)
  Change at Week 24:General health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24:General health | 1.69 (11.03) | 3.64 (10.99) | 4.70 (12.88) | 4.17 (13.82)
  Change at Week 24:Physical Function: number analyzed (Participants) | 153 | 150 | 150 | 155
  Change at Week 24:Physical Function | 6.24 (16.12) | 9.97 (16.87) | 12.99 (22.00) | 14.25 (21.60)
  Change at Week 24: Role Physical: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24: Role Physical | 7.55 (16.05) | 12.04 (20.21) | 13.88 (26.31) | 13.63 (22.54)
  Change at Week 24: Bodily Pain: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24: Bodily Pain | 9.16 (17.76) | 11.39 (18.79) | 15.91 (21.97) | 14.94 (21.55)
  Change at Week 24: Vitality: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24: Vitality | 3.77 (12.01) | 6.46 (14.63) | 6.83 (17.58) | 6.61 (15.31)
  Change at Week 24:Social Function: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24:Social Function | 3.73 (18.25) | 6.92 (19.62) | 8.83 (22.74) | 5.73 (19.60)
  Change at Week 24:Role Emotional: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24:Role Emotional | 3.30 (17.19) | 7.72 (17.80) | 7.56 (23.81) | 5.97 (22.19)
  Change at Week 24: Mental Health: number analyzed (Participants) | 154 | 150 | 150 | 155
  Change at Week 24: Mental Health | 1.40 (11.34) | 3.53 (13.01) | 1.73 (13.94) | 1.60 (15.06)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: The SF-36 health survey was a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional, domain 8= mental health. Total score for each domain are scaled 0 (minimum) to 100 (maximum), where higher score indicates highest level of functioning. These 8 domains were also summarized as summary scores: mental component aggregate (MCA) and physical component aggregate (PCA). Total score range for the each summary scores =0 to 100, where higher scores represented higher level of functioning. Higher summary scores indicated a better health related quality of life.
Time Frame: Baseline, Week 12, 24
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. BOCF method was used to impute missing values. Here, 'Overall Number of Participants Analyzed', signified number of participants evaluable for this outcome measure for respective reporting groups.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 153 | 150 | 150 | 155
Units on a scale
  Baseline: MCA | -0.03 (1.20) | 0.18 (1.15) | 0.06 (1.26) | 0.11 (1.29)
  Baseline: PCA | -1.90 (0.72) | -1.99 (0.82) | -1.96 (0.77) | -1.97 (0.76)
  Change at Week 12: MCA | 0.15 (0.73) | 0.19 (0.81) | 0.26 (1.02) | 0.10 (0.96)
  Change at Week 12: PCA | 0.29 (0.64) | 0.66 (0.90) | 0.89 (1.05) | 0.84 (1.02)
  Change at Week 24: MCA | 0.04 (0.69) | 0.20 (0.70) | 0.12 (0.88) | 0.04 (0.87)
  Change at Week 24: PCA | 0.31 (0.63) | 0.42 (0.73) | 0.60 (0.91) | 0.61 (0.86)

25. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: Intent-to-treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo).
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 155 | 155 | 154 | 157
Days | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events. | NA [NA to NA] — Median and full range cannot be estimated due to less number of participants with events.

26. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. Percentage of participants with any use of rescue medication during the particular study week were summarized.
Time Frame: Week 2, 4, 8, 12 ,16, 24
Population: mITT analysis set included all randomized participants who received at least 1 dose of intravenous study medication (either tanezumab or matching placebo), except for those who were potentially unblinded at a study site. LOCF method was used to impute missing values. Here, 'Number Analyzed', signified number of participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
Percentage of participants
  Week 2: number analyzed (Participants) | 152 | 151 | 147 | 155
  Week 2 | 46.1 | 37.1 | 36.1 | 37.4
  Week 4: number analyzed (Participants) | 153 | 151 | 148 | 156
  Week 4 | 45.8 | 26.5 | 23.6 | 23.1
  Week 8: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 8 | 30.7 | 26.5 | 22.1 | 29.5
  Week 12: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 12 | 25.5 | 22.5 | 15.4 | 20.5
  Week 16: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 16 | 23.5 | 24.5 | 24.2 | 16.7
  Week 24: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 24 | 23.5 | 25.8 | 22.8 | 24.4

27. Secondary Outcome: Duration of Rescue Medication Use
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. Number of days participant used any of the rescue medication, during the specified week were summarized.
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: All randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. LOCF method was used to impute missing values. Here, 'Number Analyzed', signified number of participants evaluable at specified time points.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 154 | 151 | 150 | 156
days
  Week 2: number analyzed (Participants) | 152 | 151 | 147 | 155
  Week 2 | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0]
  Week 4: number analyzed (Participants) | 153 | 151 | 148 | 156
  Week 4 | 2.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 8: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 8 | 1.0 [0.0 to 7.0] | 1.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 12: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 12 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 16: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 16 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]

28. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. The total dosage of acetaminophen in mg used during the specified week were summarized.
Time Frame: Week 2, 4, 8, 12, 16, 24
Population: mITT analysis set: All randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo), except those who were potentially unblinded at study site. LOCF method was used to impute missing values. Here 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 153 | 151 | 150 | 156
milligram
  Week 2: number analyzed (Participants) | 152 | 151 | 147 | 155
  Week 2 | 3917.76 (4859.09) | 3205.30 (4485.63) | 3346.94 (5405.67) | 3306.45 (4470.46)
  Week 4: number analyzed (Participants) | 153 | 151 | 148 | 156
  Week 4 | 3676.47 (4774.68) | 2437.09 (3932.47) | 2148.65 (4331.68) | 1919.87 (3183.88)
  Week 8: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 8 | 3163.40 (4984.13) | 2811.26 (5086.17) | 2372.48 (5138.01) | 2298.08 (3592.46)
  Week 12: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 12 | 2683.01 (5597.74) | 2304.64 (4477.34) | 2093.96 (5141.37) | 1910.26 (3648.90)
  Week 16: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 16 | 2366.01 (4771.42) | 2350.99 (4710.91) | 2382.55 (5197.90) | 1666.67 (3542.07)
  Week 24: number analyzed (Participants) | 153 | 151 | 149 | 156
  Week 24 | 2496.73 (5120.42) | 2274.83 (4808.22) | 2684.56 (5787.73) | 1996.79 (3717.65)

29. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 32 that were absent before treatment or that worsened relative to pretreatment state. Adverse events included both serious and all non-serious adverse events.
Time Frame: Baseline up to Week 32
Population: Safety population included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 155 | 155 | 154 | 157
Participants
  AEs | 68 | 90 | 84 | 89
  SAEs | 6 | 5 | 7 | 6

30. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 2, 4, 6, 8, 12, 16 and 24
Description: The NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. Neurologic examination assessed strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes in order to complete the NIS. The NIS is the sum of scores of over all 37 items (24 scored 0-4; 13 scored 0-2), made separately for left and right sides, giving a possible overall score range of 0 (no impairment) to 122 (severe impairment). NIS Total score range (total of both left and right sides) was 0 (no impairment) to 244 (severe impairment), where higher scores indicated increased impairment.
Time Frame: Baseline, Week 2, 4, 6, 8, 12, 16, 24
Population: Safety population included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). Here 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 155 | 155 | 154 | 157
Units on a scale
  Change at Week 2: number analyzed (Participants) | 150 | 152 | 152 | 153
  Change at Week 2 | -0.09 (1.44) | -0.22 (1.92) | -0.21 (1.03) | -0.10 (1.40)
  Change at Week 4: number analyzed (Participants) | 132 | 144 | 144 | 141
  Change at Week 4 | -0.03 (2.29) | 0.03 (2.32) | -0.38 (1.16) | -0.45 (1.52)
  Change at Week 8: number analyzed (Participants) | 123 | 133 | 137 | 137
  Change at Week 8 | -0.23 (2.04) | -0.45 (1.74) | -0.38 (1.60) | -0.35 (1.71)
  Change at Week 12: number analyzed (Participants) | 83 | 122 | 129 | 115
  Change at Week 12 | -0.23 (1.16) | -0.40 (1.96) | -0.41 (1.71) | -0.47 (1.45)
  Change at Week 16: number analyzed (Participants) | 75 | 114 | 129 | 116
  Change at Week 16 | 0.07 (1.48) | -0.33 (2.51) | -0.36 (1.63) | -0.40 (2.07)
  Change at Week 24: number analyzed (Participants) | 59 | 102 | 116 | 111
  Change at Week 24 | -0.06 (0.83) | -0.17 (1.72) | -0.46 (1.63) | -0.20 (1.59)

ADVERSE EVENTS:
Description: Participants may have experienced both nonserious and SAE during study. Cases of osteonecrosis (ON) reported in this and other studies of this program, conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Serious Adverse Events (participants affected / at risk) | 6/155 | 5/155 | 7/154 | 6/157
Other Adverse Events (participants affected / at risk) | 50/155 | 64/155 | 58/154 | 59/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Tanezumab 2.5 mg (N=155) | Tanezumab 5 mg (N=154) | Tanezumab 10 mg (N=157)
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Tanezumab 2.5 mg (N=155) | Tanezumab 5 mg (N=154) | Tanezumab 10 mg (N=157)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 5 | 3
Nausea (Gastrointestinal disorders) | 6 | 0 | 3 | 2
Oedema peripheral (General disorders) | 1 | 3 | 3 | 7
Peripheral swelling (General disorders) | 0 | 3 | 4 | 3
Bronchitis (Infections and infestations) | 2 | 5 | 3 | 3
Influenza (Infections and infestations) | 5 | 4 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 3
Sinusitis (Infections and infestations) | 1 | 2 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 7 | 10 | 10
Urinary tract infection (Infections and infestations) | 3 | 8 | 7 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 5 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 4 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 5 | 3 | 2
Liver function test abnormal (Investigations) | 1 | 0 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 4 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6 | 4 | 10
Carpal tunnel syndrome (Nervous system disorders) | 1 | 2 | 3 | 6
Headache (Nervous system disorders) | 7 | 8 | 5 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 6 | 2 | 3
Depression (Psychiatric disorders) | 4 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 2
Hypertension (Vascular disorders) | 2 | 4 | 2 | 2
Paraesthesia (Nervous system disorders) | 6 | 8 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.